CLINICAL TRIAL: NCT04396769
Title: Family Lifestyle Overweight Prevention Program-Physical Activity Only
Acronym: FLOW-PA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Houston (Other)
Collaborators: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Craig A Johnston, Associate Professor, University of Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00015671
Record Dates: First submitted 2020-05-15; First posted 2020-05-21 (Actual); Last update posted 2020-05-22 (Actual); Status verified 2020-05

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FLOW-PA (Experimental): Participants received the physical activity component of FLOW five days a week during participants' 45-minute long physical education (PE) class period for six months. Intervention activities were designed to promote moderate-vigorous physical activity through circuit-based stations with both aerobic and strength exercises. Trained research staff partnered with PE teachers to facilitate lessons and undergraduate college students were trained to complete activities with participants.
  Interventions: Behavioral: FLOW-PA
- PE class as usual (Active Comparator): Participants had PE class as usual 5 days a week for 45 minutes.
  Interventions: Behavioral: PE class as usual

INTERVENTIONS:
Behavioral: FLOW-PA — Classes were designed to provide the opportunity to be physically activity at a moderate-vigorous level. Each station included exercise options to accommodate varying fitness levels and offer students choice. Heart rate monitors provided consistent biofeedback to students throughout the intervention. Participants were evaluated based on the number of minutes they spent each class between 60-80% of their maximal heart rate. Games were intermixed either as a station or as a break in the circuit (e.g. short game of tag half-way through the workout) to make physical activity enjoyable and engaging.
  Arms: FLOW-PA
Behavioral: PE class as usual — PE teachers were instructed to teach class as usual. Research staff were not involved in class activities or instruction. In this school district PE class as usual includes sports-based instruction in which students learn the rules to games and then practice playing.
  Arms: PE class as usual

SUMMARY:
This randomized control trial evaluates the physical activity component of the Family Lifestyle Overweight Prevention Program compared to physical education class as usual among Hispanic middle school students.

DETAILED DESCRIPTION:
Family Lifestyle Overweight Prevention Program (FLOW) is an intensive, multi-component obesity intervention designed to take place during physical education class. This intervention has established efficacy at improving standardized BMI among low income, Hispanic middle school students with overweight classification or obesity. However, the efficacy of individual components of the intervention have not been investigated. The purpose of this study was to compare only the physical activity component of FLOW to a physical education class as usual. The primary outcome of the study is time spent in moderate-vigorous physical activity. Secondarily the study evaluated the impact of the intervention on standardized BMI.

ELIGIBILITY:
Inclusion Criteria:

* age 10-17 years old
* enrolled in a middle school PE class at YES Prep Brays Oaks

Exclusion Criteria:

* pregnant
* cognitive impairment significantly below average age or grade level

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 491 (Actual)
Dates: Start 2011-08-15 (Actual); Primary Completion 2014-06-01 (Actual); Study Completion 2014-06-01 (Actual)

PRIMARY OUTCOMES:
Weekday moderate-vigorous physical activity (MVPA) | six months
  weekday (Monday-Friday) minutes/day of MVPA over time assessed with accelerometry

SECONDARY OUTCOMES:
Weekend moderate-vigorous physical activity (MVPA) | six months
  Weekend (Saturday-Sunday) minutes/day of MVPA over time assessed with accelerometry
standardized BMI (zBMI) | six months
  standardized BMI over time

CONTACTS AND LOCATIONS:
Overall Officials: Craig A Johnston, PhD, Principal Investigator — University of Houston

IPD SHARING:
Plan to Share IPD: No